CLINICAL TRIAL: NCT00810043
Title: Study of Curette Use for Obtaining Restoration of Vertebral Body Anatomy in Balloon Kyphoplasty
Brief Title: Medtronic SCORE Study - Study of Curette Use for Obtaining Restoration of Vertebral Body Anatomy in Balloon Kyphoplasty
Acronym: MDTSCORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0801 - SCORE
Record Dates: First submitted 2008-12-12; First posted 2008-12-17 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2014-04

CONDITIONS: Vertebral Body Compression Fractures (VCFs)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curette-First (Active Comparator): All of patients in the study were treated with Balloon Kyphoplasty. During Balloon Kyphoplasty, two inflatable bone tamps (IBTs) are placed into the vertebral body bilaterally via a transpedicular or extrapedicular approach under fluoroscopic guidance. In this arm, curettage was performed prior to use of inflatable bone tamps.
  Interventions: Device: Kyphon® Curette
- IBT-First (Active Comparator): All of patients in the study were treated with Balloon Kyphoplasty. During Balloon Kyphoplasty, two inflatable bone tamps (IBTs) are placed into the vertebral body bilaterally via a transpedicular or extrapedicular approach under fluoroscopic guidance. In this arm, inflatable bone tamps were used prior to curettage, then followed by a second inflation of the bone tamps.
  Interventions: Device: Kyphon® Curette

INTERVENTIONS:
Device: Kyphon® Curette — The Kyphon® Curette is intended to scrape and score bone in the spine. It may be used as an adjunctive device with Kyphon's family of standard access and fracture reduction instruments designed to treat compression fracture during balloon kyphoplasty procedures

SUMMARY:
The objective of this study is to measure the effect that the scraping and scoring of vertebral cancellous bone using the Kyphon® Curette has on vertebral body anatomy height restoration and angular deformity correction during a balloon kyphoplasty procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 50 years
* One painful VCF meeting all of the following criteria:

  * Fracture due to diagnosed or suspected underlying primary or secondary osteoporosis
  * VCF is between T5 and L5
  * VCF shows hyperintense signal on STIR or T2 weighted MRI
  * VCF has at least 15% height loss as visualized on plain radiograph
  * Identified painful VCF has at least superior and one normal vertebrae within 2 levels inferior.
  * Either the immediate superior OR the immediate inferior vertebral body (but not both) may have a chronic fracture that does not need treatment.
* Patient states availability for all study visits
* Patient is able to understand the risks and benefits of participating in the study and is willing to provide written informed consent

Exclusion Criteria:

* Patient is unable to undergo MRI
* Patient shows evidence of edema in vertebral bodies other than index level on MRI
* Patient is unable to stand for pre-operative and post-operative x-rays
* Patient body mass index (BMI) is greater than 35 kg/m2
* Patient is pregnant, or of child-bearing potential and not using contraception
* Vertebral body (VB) morphology or configuration is such that balloon kyphoplasty is not technically feasible or clinically appropriate for the index VCF
* Index fracture is result of high-energy trauma
* Suspected or proven cancer inside any VB
* Disabling back pain due to causes other than acute fracture
* Spine stabilization beyond balloon kyphoplasty required for index VCF
* Pre-existing conditions contrary to balloon kyphoplasty, such as:

  * Irreversible coagulopathy or bleeding disorder. Note that patients on Coumadin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and re-initiation of anticoagulants.
  * Allergy to any device materials (e.g., bone cement) for balloon kyphoplasty. Note that in patients with allergy to iodine-based contrast, other marketed approved non-iodine contrast solutions may be used.
  * Any evidence of VB or systemic infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Fueredi, M.D., Principal Investigator — Aurora Heath Care, Inc.
Locations (13):
- United States (3):
  - Foundation for Orthopaedic Research and Education, Temple Terrace, Florida
  - Atrium Medical Center, Middletown, Ohio
  - Aurora Medical Group, Memorial Hospital of Burlington, Burlington, Wisconsin
- Belgium (2):
  - CHC - Les Cliniques Saint-Joseph, Liège
  - St. Augustinus ziekenhuis, Wilrijk
- Germany (8):
  - Charité Campus Virchow-Klinikum Berlin, Berlin
  - Kliniken im Naturpark Altmühltal, Eichstätt
  - Klinikum Kempten, Kempten
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Paracelcus-Klinik München, München
  - Kliniken Dr. Erler, Nuremberg
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
  - Asklepios Orthopadische Klinik Lindenlohe, Schwandorf in Bayern

REFERENCES:
- [Derived] Bastian L, Schils F, Tillman JB, Fueredi G; SCORE Investigators. A randomized trial comparing 2 techniques of balloon kyphoplasty and curette use for obtaining vertebral body height restoration and angular-deformity correction in vertebral compression fractures due to osteoporosis. AJNR Am J Neuroradiol. 2013 Mar;34(3):666-75. doi: 10.3174/ajnr.A3363. Epub 2012 Nov 22. PMID 23179647

RESULTS

PARTICIPANT FLOW:
Groups:
- Curette-First: Use of the curette prior to use of the inflatable bone tamps
- IBT-First: Use of the inflatable bone tamps prior to using the curette
- Non-treated Patients: Patients who met the enrollment criteria at screening who had terminated prior to surgery or those who no longer met the inclusion criteria due to new fractures prior to surgery. These patients were never randomized to treatment because randomization was performed in the operating room.
Period: Overall Study
Arm/Group | Curette-First | IBT-First | Non-treated Patients
Started | 57 | 55 | 8
Completed | 53 | 54 | 0
Not Completed | 4 | 1 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Death | 2 | 0 | 0
Not completed — Unrelated medical problem | 0 | 1 | 0
Not completed — Non-medical problem | 0 | 0 | 1
Not completed — No longer met enrollment criteria | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curette-First | IBT-First | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (8.4) | 76.0 (9.4) | 74.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 10 | 14 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 55 | 55 | 110
  Hispanic | 1 | 0 | 1
  Middle Eastern | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 31
  Belgium | 18 | 16 | 34
  Germany | 26 | 21 | 47
Smoking history [Number; unit: Participants]
  Never Smoked | 36 | 36 | 72
  Current Smoker | 7 | 5 | 12
  Former Smoker | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Absolute Vertebral Body Height Restoration as a Percent (Post-procedure Change From Baseline)
Time Frame: Baseline and 48-hr post-procedure
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Curette-First: Use of curette prior to use of inflatable bone tamps
- IBT-First: Use of inflatable bone tamps prior to use of the curette, followed by inflatable bone tamps
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
percent change
  Anterior vertebral measurement (n=52, 50) | 9.72 (12.85) [6.1 to 13.3] | 11.77 (13.23) [8.0 to 15.5]
  Mid-vertebral measurement (n=52, 50) | 8.14 (9.96) [5.4 to 10.9] | 9.07 (10.31) [6.1 to 12.0]
  Posterior vertebral measurement (n=52, 50) | 2.59 (5.15) [1.2 to 4.0] | 4.21 (6.49) [2.4 to 6.1]
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Anterior vertebral body height restoration as a percent (Post-procedure change from baseline); Test type: Superiority or Other; p = 0.430, t-test, 2 sided
Statistical Analysis 2: Comparison: Curette-First vs IBT-First; Middle vertebral body height restoration as a percent (Post-procedure change from baseline); Test type: Superiority or Other; p = 0.643, t-test, 2 sided
Statistical Analysis 3: Comparison: Curette-First vs IBT-First; Posterior vertebral body height restoration as a percent (Post-procedure change from baseline); Test type: Superiority or Other; p = 0.165, t-test, 2 sided

2. Secondary Outcome: Index Vertebral Body Height Restored in Millimeters.
Description: Vertebral Body Height (VBH) was measured at anterior, midpoint, and posterior of index vertebral bodies. The data presented is the absolute height restored (AHR) between two time points.
Time Frame: Baseline and 48 hours after procedure
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
mm
  Anterior VBH at baseline (n=54, 53) | 14.15 (5.25) | 14.27 (5.02)
  Anterior VBH at 48 hr post-procedure (n=56, 51) | 16.65 (4.75) | 17.32 (4.33)
  Anterior change in VBH (n=53, 50) | 2.28 (2.89) | 2.78 (3.11)
  Midpoint VBH at baseline (n=54, 53) | 13.98 (4.12) | 14.21 (4.07)
  Midpoint VBH at 48 hr post-procedure (n=56, 51) | 16.22 (4.01) | 16.62 (3.39)
  Midpoint change in VBH (n=53, 50) | 1.98 (2.38) | 2.25 (2.58)
  Posterior VBH at baseline (n=54, 53) | 22.79 (3.61) | 22.94 (4.32)
  Posterior VBH at 48 hr post-procedure (n=56, 51) | 23.57 (3.99) | 24.02 (3.59)
  Posterior change in VBH (n=53, 50) | 0.65 (1.29) | 1.05 (1.65)
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Anterior VBH restored; Test type: Superiority or Other; p = 0.402, t-test, 2 sided
Statistical Analysis 2: Comparison: Curette-First vs IBT-First; Middle VBH restored; Test type: Superiority or Other; p = 0.578, t-test, 2 sided
Statistical Analysis 3: Comparison: Curette-First vs IBT-First; Posterior VBH restored; Test type: Superiority or Other; p = 0.166, t-test, 2 sided

3. Secondary Outcome: Amount of Vertebral Body Height (VBH) Gained From IBTs Alone
Description: Since all patients were treated in the prone position with chest and hip bolsters (this is referred to as postural reduction), vertebral body height (VBH) gained from IBTs alone was reported as the change of vertebral body height measured intra-operatively after postural reduction with bolsters to the 1st round of IBT inflation.
Time Frame: Intra-operative measurement after postural reduction with Bolsters and intra-operative measurement after 1st round of IBT inflation.
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | IBT-First
Number analyzed (Participants) | 55
mm
  Anterior VBH at intra-op with Bolster (n=47) | 17.03 (4.72)
  Anterior VBH at Intra-op 1st IBT (n=49) | 18.40 (4.67)
  Anterior VBH change (n=47) | 1.25 (1.94)
  Middle VBH at intra-op with Bolster (n=47) | 15.99 (3.60)
  Middle VBH at Intra-op 1st IBT (n=49) | 17.00 (3.32)
  Middle VBH change (n=47) | 0.94 (1.38)
  Posterior VBH at intra-op with Bolster (n=47) | 23.68 (3.85)
  Posterior VBH at Intra-op 1st IBT (n=49) | 24.05 (3.61)
  Posterior VBH change (n=47) | 0.37 (0.81)

4. Secondary Outcome: Amount of Vertebra Body Height (VBH) Gained by Postural Reduction
Time Frame: baseline and intra-operative
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
mm
  Anterior VBH at baseline (n=54, 53) | 14.15 (5.25) | 14.27 (5.02)
  Anterior VBH at intra-op with Bolster (n=50, 47) | 16.93 (4.99) | 17.03 (4.72)
  Anterior VBH gained (n=47, 46) | 2.96 (3.55) | 3.05 (3.21)
  Middle VBH at baseline (n=54, 53) | 13.98 (4.12) | 14.21 (4.07)
  Middle VBH at intra-op with Bolster (n=50, 47) | 15.96 (4.36) | 15.99 (3.60)
  Middle VBH gained (n=47, 46) | 1.88 (2.64) | 2.14 (2.48)
  Posterior VBH at baseline (n=54, 53) | 22.79 (3.61) | 22.94 (4.32)
  Posterior VBH at Intra-op with Bolser (n=50, 47) | 23.41 (4.02) | 23.68 (3.85)
  Posterior VBH gained (47, 46) | 0.64 (1.69) | 0.95 (1.53)
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Anterior VBH gained by postural reduction; Test type: Superiority or Other; p = 0.900, t-test, 2 sided
Statistical Analysis 2: Comparison: Curette-First vs IBT-First; Middle VBH gained by postural reduction; Test type: Superiority or Other; p = 0.620, t-test, 2 sided
Statistical Analysis 3: Comparison: Curette-First vs IBT-First; Posterior VBH gained by postural reduction; Test type: Superiority or Other; p = 0.349, t-test, 2 sided

5. Secondary Outcome: Deformity Correction Assessed by Vertebral Body Kyphosis Angle (VBA)
Description: The vertebral body kyphosis angle (VBA) was defined as the angle formed by lines drawn parallel to the caudal and cranial fractured vertebral body endplates. Correction of angular deformity was expressed as a difference of absolute values between pre- and post-operative values. Any positive change indicated an improvement of angular correction and was defined as a change in angulation toward 0 degrees. Any negative change indicated a worsening of angular correction, and is defined as a change away from 0 degrees.
Time Frame: Baseline and 48 hr post-procedure
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
degree
  VBA at baseline (n=54, 53) | -15.5 (7.17) | -15.1 (7.82)
  VBA at 48 hr post-procedure (n=56, 51) | -12.4 (6.23) | -11.5 (6.84)
  Angle change (n=53, 50) | 2.88 (4.48) | 3.00 (4.42)
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Test type: Superiority or Other; p = 0.889, t-test, 2 sided

6. Secondary Outcome: Deformity Correction Assessed by Local Cobb Angle (LCA)
Description: The local Cobb angle (LCA) was defined as the angle formed by lines drawn parallel to the superior endplate of the vertebral body above and the inferior endplate of the vertebral body below. Correction of angular deformity was expressed as a difference of absolute values between pre- and post-operative values. Any positive change indicated an improvement of angular correction and was defined as a change in angulation toward 0 degrees. Any negative change indicated a worsening of angular correction, and is defined as a change away from 0 degrees.
Time Frame: baseline and 48 hr post-procedure
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
degree
  LCA at Baseline (n=53, 50) | -13.8 (15.09) | -11.5 (17.82)
  LCA at 48 hr post-procedure (n=56, 49) | -10.70 (16.28) | -7.88 (16.29)
  Angle change (n=52, 48) | 1.36 (3.68) | 1.87 (3.63)
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Test type: Superiority or Other; p = 0.486, t-test, 2 sided

7. Secondary Outcome: Change in Back Pain.
Description: Back pain was assessed by a numeric rating scale (Scale 1-10), with higher scores denoting worse pain.
Time Frame: Baseline and 48 hr post-procedure
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
units on a scale
  Back pain at baseline (n=57, 55) | 7.7 (1.3) | 7.5 (1.3)
  Back pain at 48 hr post-procedure (n=57, 55) | 3.0 (2.0) | 3.3 (1.9)
  Back pain change from baseline (n=57, 55) | -4.7 (1.9) | -4.2 (1.9)
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Test type: Superiority or Other; p = 0.144, t-test, 2 sided

8. Secondary Outcome: Change in Ambulatory Status
Description: Ambulatory status was assessed by subjective patient questionnaire.
Time Frame: Baseline and 48 hrs post-procedure
Population: Modified intention to treat - all randomized patients who received balloon kyphoplasty treatment.
Measure: Number; unit: participants
Arm/Group | Curette-First | IBT-First
Number analyzed (Participants) | 57 | 55
participants
  Able to walk without assistance -- baseline | 36 | 34
  Able to walk with aid -- baseline | 18 | 21
  Must use wheelchair or bedridden -- baseline | 3 | 0
  Able to walk without assistance -- 48 hrs post-op | 48 | 42
  Able to walk with aid -- 48 hrs post-op | 9 | 12
  Must use wheelchair or bedridden -- 48 hrs post-op | 0 | 1
  No change | 43 | 40
  Improved | 13 | 11
  Worsened | 1 | 4
Statistical Analysis 1: Comparison: Curette-First vs IBT-First; Test type: Superiority or Other; p = 0.360, Chi-squared

ADVERSE EVENTS:
Arm/Group | Curette-First | IBT-First
Serious Adverse Events (participants affected / at risk) | 5/57 | 8/55
Other Adverse Events (participants affected / at risk) | 12/57 | 11/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curette-First (N=57) | IBT-First (N=55)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curette-First (N=57) | IBT-First (N=55)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Procedural vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion postoperative (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less